CLINICAL TRIAL: NCT00533910
Title: Effect of Rifaximin on Driving Performance, Psychometric Test Performance and Quality of Life in Cirrhotic Patients With Minimal Hepatic Encephalopathy: Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Rifaximin in Minimal Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Jasmohan Bajaj, Associate Professor of Medicine, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00006863
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hepatic Encephalopathy
Keywords: Minimal hepatic encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Will be given placebo and follow the exact procedures as the experimental section
  Interventions: Drug: placebo
- Drug (Experimental)
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — 550mg BID rifaximin for 8 weeks
  Arms: Drug
Drug: placebo — same as the experimental arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether alteration of gut flora with rifaximin can lead to improvement in driving performance, psychometric test performance, and quality of life in patients with minimal hepatic encephalopathy (MHE) and cirrhosis in a randomized, blinded, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Cirrhosis diagnosed on clinical grounds
* MHE diagnosed by abnormalities in a psychometric battery (NCT-A, NCT-B, ICT BDT and DST impaired beyond 2 standard deviations of known control values on any of the above 3 tests will be considered to have MHE)
* Current drivers (valid driving license and driving at least 20 miles/week)
* All women of child-bearing potential will be required to use effective contraception

Exclusion Criteria:

* Current or recent (< 6 month) use of alcohol (AUDIT questionnaire will be used; any cirrhotic with a value of > 0 will be excluded) and a positive blood alcohol level
* Use of antibiotics within last 6 weeks
* Allergy to rifaximin, rifabutin, rifampin, or rifapentine
* Infection or gastrointestinal hemorrhage within the last 6 weeks
* Renal insufficiency
* Hepatocellular carcinoma
* Psychoactive drug use, including interferon concurrently
* Non-drivers and those who drive less than 20 miles/week
* Pregnancy and breastfeeding
* Excluding patients with OHE:

  * Detailed neurological examination to check for dysarthria, asterixis, ataxia and disorientation
  * Detailed history-taking from friends/relatives only after taking the patient's permission
  * Mini-mental status examination > 25
  * Episode of overt (clinical hepatic encephalopathy) within 6 months
  * Current treatment with lactulose, rifaximin, zinc, or metronidazole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MBBS, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Bajaj JS, Heuman DM, Wade JB, Gibson DP, Saeian K, Wegelin JA, Hafeezullah M, Bell DE, Sterling RK, Stravitz RT, Fuchs M, Luketic V, Sanyal AJ. Rifaximin improves driving simulator performance in a randomized trial of patients with minimal hepatic encephalopathy. Gastroenterology. 2011 Feb;140(2):478-487.e1. doi: 10.1053/j.gastro.2010.08.061. Epub 2010 Sep 21. PMID 20849805
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rifaximin
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rifaximin | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Driving Performance
Description: Total driving errors at the end of drug/placebo. Minimum is zero, maximum is not defined. Higher number indicates greater errors.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: raw number of driving errors
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 21 | 21
raw number of driving errors | 7.6 (3.9) | 5.5 (3.8)

2. Secondary Outcome: Psychometric Test Performance
Description: Z score of combined cognitive tests at end of rifaximin/placebo; higher scores indicate better psychometric test performance
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Z scores
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 21 | 21
Z scores | 0.46 (0.17) | 1.19 (0.24)

3. Secondary Outcome: Total Sickness Impact Profile Score
Description: Total score ranging from 0 through >100 at the end of drug/placebo. Higher score indicates worse QOL
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 21 | 21
score on a scale | 12 (3) | 10 (2)

ADVERSE EVENTS:
Time Frame: 8 weels
Description: Same as the ones in www.clinicaltrials.gov definitions
Arm/Group | Placebo | Rifaximin
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No